CLINICAL TRIAL: NCT06469190
Title: An Exploratory Clinical Study of the Safety and Efficacy of Anti-CD19 Chimeric Antigen Receptor NK Cell Injections (KN5501) in the Treatment of Relapsed/Refractory Immune Nephropathy
Brief Title: An Exploratory Clinical Study of Anti-CD19 CAR NK Cell (KN5501) in the Treatment of Relapsed/Refractory Immune Nephropathy
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Changhai Hospital (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHEC2024-188
Record Dates: First submitted 2024-06-17; First posted 2024-06-21 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2024-07

CONDITIONS: Nephropathy
MeSH Terms: conditions — Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- KN5501 (Experimental)
  Interventions: Biological: anti-CD19 CAR NK cells

INTERVENTIONS:
Biological: anti-CD19 CAR NK cells — Patients will receive Fludarabine (30 mg/m2 per day) and Cyclophosphamide (300mg/m2 per day) on day -5, -4, and -3. Multiple doses of anti-CD19 CAR NK cells (KN5501) will infused in each group using the "3 + 3" dose-escalation strategy.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and effectiveness of anti-CD19 CAR NK cell injection (KN5501) in patients with immune nephropathy. 36 patients are planned to be enrolled in the dose-escalation trial. The primary endpoints are DLT and TEAEs. The secondary endpoints are the overall response rates (ORR) and disease control rate (DCR)

ELIGIBILITY:
Common Inclusion Criteria:

1. Age: ≥ 18 years old and ≤ 70 years old, male or female;
2. Positive CD19 expression in peripheral blood B cells as determined by flow cytometry;
3. The functions of important organs meet the following requirements:

   1. Bone marrow hematopoietic function: a. White blood cell count ≥ 3 x 10^9/L b. Neutrophil count ≥ 1 x 10^9/L (no colony-stimulating factor treatment within 2 weeks before examination); c. Hemoglobin ≥60g/L.
   2. Liver function: ALT ≤ 3 x ULN,AST≤3 x ULN, TBIL≤1.5 x ULN(excluding Gilbert syndrome, total bilirubin ≤ 3.0 x ULN)
   3. Coagulation function: International standardized ratio (INR) ≤ 1.5 x ULN, prothrombin time (PT) ≤1.5 x ULN.
   4. Cardiac function: good hemodynamic stability, left ventricular ejection fraction (LVEF) ≥55%.
4. Female subjects of childbearing potential and male subjects whose partner is a female of childbearing potential are required to use medically approved contraception or abstain from sex for at least 6 months during and at least 6 months after the end of the study treatment period; female subjects of childbearing potential have had a negative serum HCG test within 7 days prior to study enrollment and are not lactating;
5. Voluntarily participate in this clinical study, sign an informed consent form, have good compliance, and cooperate with follow-up.

Criteria for Recurrent/refractory primary membranous nephropathy

1. Primary membranous nephropathy diagnosed pathologically by renal biopsy;
2. Screening period 24-hour urine protein quantification ≥3.5 g;
3. Individuals who have not achieved partial remission (PR) after more than 6 months of treatment with hormonal and/or cytotoxic drugs, immunosuppressive therapy, and/or biologics (including but not limited to anti-CD20 monoclonal antibody); or individuals who have relapsed again after achieving complete remission/partial remission (CR/PR) with treatment (24h urine protein quantification ≥3.5g);
4. Glomerular filtration rate (eGFR, CKD-EPI formula) ≥45 ml/min/1.73m2 during the screening period.

Criteria for Relapsed/refractory IgA nephropathy

1. Primary IgA nephropathy pathologically confirmed by renal biopsy;
2. Treated (ACEI/ARB analogs) for at least 3 months;
3. Treatment with hormonal and/or cytotoxic drugs, immunosuppressive therapy, and/or biologics (including, but not limited to anti-CD20 monoclonal antibody) for more than 6 months, 24-hour urine protein quantification ≥ 1.0 g; or rapid progression of renal function (≥ 50% decrease in eGFR within 3 months); or relapse after treatment to achieve complete remission/partial remission (CR/PR) (24-hour urine protein quantification ≥ 1.0 g);
4. Glomerular filtration rate (eGFR, CKD-EPI formula) ≥30 ml/min/1.73m2 during the screening period.

Criteria for Relapsed/refractory ANCA-associated vasculitis

1. Meets 2022 ACR/EULAR diagnostic criteria for ANCA vasculitis, including microscopic polyangiitis, granulomatous polyangiitis, eosinophilic granulomatous polyangiitis;
2. Positive ANCA related antibodies (MPO-ANCA or PR3-ANCA positive);
3. Renal biopsy pathology consistent with renal damage in ANCA-associated vasculitis;
4. The Birmingham Vasculitis Activity Scale (BVAS) is ≥ 15 points (a total score of 63 points), indicating the activity of the vasculitis condition;
5. BVAS score includes at least 2 abnormalities in the renal program;
6. Definition of relapse/refractory : ineffective conventional treatment or relapse of disease activity after remission. Definition of routine treatment: use of glucocorticoids (more than 1 mg/kg/d) and cyclophosphamide for ≥3 months, and any of the following immunomodulatory drugs: antimalarial drugs, azathioprine, mycophenolate mofetil, methotrexate, leflunomide, tacrolimus, cyclosporine, as well as biological agents such as rituximab and belimumab;
7. Glomerular filtration rate (eGFR, CKD-EPI formula) ≥15 ml/min/1.73m2 during the screening period.

Common exclusion Criteria:

1. Individuals with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, tozumabs), or subjects with a history of severe allergic reactions;
2. Existence or suspicion of uncontrollable or treatable fungal, bacterial, viral or other infections;
3. Individuals with central nervous system disorders caused by ADs or not caused by ADs (including epilepsy, psychiatric disorders, organic encephalopathy syndromes, cerebrovascular accidents, encephalitis, central nervous system vasculitis);
4. Individuals with relatively serious heart diseases, such as angina pectoris, myocardial infarction, heart failure, and arrhythmia;
5. Subjects with congenital immunoglobulin deficiency;
6. Subjects with malignant tumors (except for non-melanoma skin cancer and in situ cervical, bladder, and breast cancers that have been disease-free for more than 5 years);
7. Subjects with end-stage renal failure;
8. Subjects with positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) and HBV DNA titer in peripheral blood higher than the upper limit of detection; Patients with positive hepatitis C virus (HCV) antibodies and positive peripheral blood HCV RNA; People who are positive for human immunodeficiency virus (HIV) antibodies; Those who have tested positive for syphilis;
9. Subjects with mental illness and severe cognitive impairment;
10. Subjects who have received other clinical trial treatment within 3 months;
11. Pregnant or intending to conceive women;
12. In the opinion of the investigator, there are other reasons why subjects cannot be included in this study.

Exclusion Criteria for Recurrent/refractory primary membranous nephropathy

1. Secondary membranous nephropathy (e.g., hepatitis B, systemic lupus erythematosus, drug-associated, malignancy-associated, etc.), or in combination with other renal diseases confirmed by renal biopsy;
2. Type 1 or type 2 diabetes.

Exclusion Criteria for Relapsed/refractory IgA nephropathy

1. Exclude secondary IgA nephropathy, including but not limited to: anaphylactic purpura, ankylosing spondylitis, systemic lupus erythematosus, desiccation syndrome, viral hepatitis, cirrhosis of the liver, rheumatoid arthritis, and mixed connective tissue disease; or in combination with other renal diseases confirmed by renal biopsy;
2. Crescentic nephritis (pathologic diagnosis of >50% crescentic bodies), micrognathic nephropathy with IgA deposition, and other specific types of pathologic or clinical renal disease.

Exclusion Criteria for Relapsed/refractory ANCA-associated vasculitis

1. Estimated glomerular filtration rate (eGFR) <15 mL/min/1.73 m2;
2. If the patient has alveolar hemorrhage invasive lung ventilation is required, estimated to last longer than the screening period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-06-21 (Actual); Primary Completion 2025-06-20 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-Limiting Toxicity (DLT) | up to 48 weeks after infusion
  To characterize the safety of anti-CD19 CAR NK Cells (KN5501) for Relapsed/Refractory Immune Nephropathy
Incidence of Treatment Emergent Adverse Events (TEAEs) | up to 48 weeks after infusion
  To characterize the safety of anti-CD19 CAR NK Cells (KN5501) for Relapsed/Refractory Immune Nephropathy

SECONDARY OUTCOMES:
The overall response rate (ORR) | 1, 3, 6, 12 and 12 months after infusion
  To characterize the efficacy of anti-CD19 CAR NK Cell Therapy for Relapsed/Refractory Immune Nephropathy
Disease control rate (DCR) | 1, 3, 6, 12 and 12 months after infusion
  To characterize the efficacy of anti-CD19 CAR NK Cell Therapy for Relapsed/Refractory Immune Nephropathy
B cell depletion rate | 1, 3, 6, 12 and 12 months after infusion
  To characterize the efficacy of anti-CD19 CAR NK Cell Therapy for Relapsed/Refractory Immune Nephropathy
B cell reconstitution | 1, 3, 6, 12 and 12 months after infusion
  To characterize the efficacy of anti-CD19 CAR NK Cell Therapy for Relapsed/Refractory Immune Nephropathy

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changhai hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No